CLINICAL TRIAL: NCT02738437
Title: Kryptonite - a Novel Osteosynthesis Method for Median Sternotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Rikke Vestergaard, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Kryptonite
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: osteogenesis; Positron-Emission Tomography; Radiostereometric analysis
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Control Group receiving standard treatment
- intervention group (Active Comparator): Intervention Group receiving the standard treatment and the kryptonite-bone cement
  Interventions: Device: Kryptonite-bone cement

INTERVENTIONS:
Device: Kryptonite-bone cement
  Arms: intervention group

SUMMARY:
The aim of this study was to investigate the beneficial effect of bone cement in combination with wire cerclage on the stability of the sternum following median sternotomy.

One half of the patients received only wire cerclage the other both bone cement and wire cerclage.

DETAILED DESCRIPTION:
The aim of this study was to investigate the beneficial effect of bone cement in combination with wire cerclage on the stability of the sternum following median sternotomy.

It has been shown previously that wire cerclage alone does not provide a stabile osteosynthesis following median sternotomy. The hypothesis is that if a stabile osteosynthesis can be achieved patient recovery can be hastened and patient discomfort and pain reduced.

One half of the patients received only wire cerclage the other both bone cement and wire cerclage.

The stability of the sternum was evaluated using radiostereometric analysis, PET-CT and patient reported outcomes in the form of SF-36 and VAS.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective Heart surgery

Exclusion Criteria:

* none

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Radiostereometric analysis | 6 weeks, 3 and 6 months
  Evaluation of change of Stability/mobility of the osteotomy evaluated using radiostereometric analysis. The distance in cm between sternal halves is measured.
Evaluation of sternal healing using PET-scan | 3 and 6 months
  Change in bone healing using PET-scan

SECONDARY OUTCOMES:
Pain | 3 weeks, 3 and 6 months
  evaluation of the patients pain-levels using VAS
General well-being | 3 weeks, 3 and 6 months
  evaluation of the patients general well-being using SF-36
sternal discomfort | 3 weeks, 3 and 6 months
  evaluation of the specific discomfort related to median sternotomy using a specific questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Skejby, Dept. of Cardiothoracic surgery, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Vestergaard RF, Soballe K, Hasenkam JM, Stilling M. Sternal instability measured with radiostereometric analysis. A study of method feasibility, accuracy and precision. J Cardiothorac Surg. 2018 May 18;13(1):41. doi: 10.1186/s13019-018-0735-4. PMID 29776382